CLINICAL TRIAL: NCT04562896
Title: Iterative Design of Custom Dynamic Orthoses to Reduce Articular Contact Stress
Acronym: PRMRP-FPA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: University of Delaware (Other); Bio-Mechanical Composites (Unknown); Fabtech Systems (Unknown)
Responsible Party: Principal Investigator, Jason Wilken, Director of Collaborative Research and Development, Associate Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 202002769; CDMRP-PR172087 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-08-31; First posted 2020-09-24 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-04

CONDITIONS: Ankle Fractures; Post-traumatic Osteoarthritis; Osteoarthritis Ankle
Keywords: Carbon Fiber; Gait Analysis; Ankle Foot Orthosis; Arthritis; Biomechanics; Ankle; Adult
MeSH Terms: conditions — Ankle Fractures; Arthritis

STUDY DESIGN:
Intervention Model Description: All participants will be cast and fit with three carbon fiber custom dynamic orthoses (CDOs). Each CDO will differ from the others in design and will be labeled as CDO-A, CDO-B and CDO-C. Participants will be randomly assigned to one of six CDO testing sequences (ABC, ACB, BCA, BAC, CAB, CBA) to prevent testing order from influencing study results. Multiple rounds of evaluation (~5 rounds) with small groups of participants in each round (n=~6) will be used.
Who Masked: Participant
Masking Description: Participants will be blinded to the different design variations of each device, and will only be introduced to each device as CDO-A, CDO-B or CDO-C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- No Device (No Intervention): Participants will be evaluated without a CDO.
- CDO-A (Experimental): The first design variant will be designated CDO-A
  Interventions: Device: Custom Carbon Fiber Dynamic Orthosis (CDO)
- CDO-B (Experimental): The second design variant will be designated CDO-B
  Interventions: Device: Custom Carbon Fiber Dynamic Orthosis (CDO)
- CDO-C (Experimental): The third design variant will be designated CDO-C
  Interventions: Device: Custom Carbon Fiber Dynamic Orthosis (CDO)

INTERVENTIONS:
Device: Custom Carbon Fiber Dynamic Orthosis (CDO) — The custom carbon fiber dynamic orthoses will consist of a semi-rigid foot plate, a posterior carbon fiber strut, and a proximal cuff below the knee.
  Other Names: Ankle Foot Orthosis
  Arms: CDO-A; CDO-B; CDO-C

SUMMARY:
The proposed study evaluates the effect of carbon fiber brace design on forces across the ankle joint. Research suggests that ankle arthritis develops after ankle fracture, in part, due to elevated forces on the cartilage. It is expected that carbon fiber braces can be designed to reduce forces in the ankle joint and thereby reduce the risk of developing arthritis following traumatic injury. In this study, brace geometry will be varied to determine how these changes influence the forces experienced by ankle cartilage. The proposed study will provide evidence that can be used by clinicians and researchers to design braces that most effectively reduce forces on ankle cartilage.

DETAILED DESCRIPTION:
The primary purpose of this line of research is to investigate the effects of carbon fiber custom dynamic orthosis (CDO) design on the forces and contact stress at the ankle, with the goal of reducing the development of post traumatic osteoarthritis (PTOA) in the ankle. Research suggests that ankle arthritis develops, in part, due to increased contact stresses within the ankle joint following fracture. It is expected that reducing articular contact stress at the ankle has the potential to delay or prevent the development of PTOA. CDOs have been shown to significantly improve function following extremity injury, and show promise for offloading the injured limb after severe lower extremity injuries. Therefore, the proposed effort is designed to evaluate how different CDO design factors influence offloading and therefore the reduction of forces and articular contact stress at the ankle.

Adult participants will be evaluated while wearing carbon fiber braces of varied geometry. The primary dependent measure is ankle joint contact stress. Following consent and enrollment computerized tomography (CT) images will be used to determine the geometry of the joint articular surfaces. Ankle contact stress will be calculated using discrete element analysis and biomechanical data collected in subsequent data collection.

Participants will be cast and fit for three CDOs with varied geometry. Participants will be blinded to the design variation of each device and will only know them as CDO-A, CDO-B, or CDO-C. Testing will be completed under 4 conditions: No-CDO, CDO-A, CDO-B, CDO-C, with each bracing condition (A/B/C) representing a CDO design variant. Physical performance measures will incorporate tests of agility, speed, and lower limb power to ensure that changes to device design do not negatively affect physical function. Questionnaires will be used to evaluate participants' current and desired activity level, pain with and without CDO use, satisfaction with the devices, perception of comfort and smoothness between devices, and preference between CDOs. Semi-structured interviews will be completed to fully capture the participant's perspective. Lower limb forces and motion will be assessed using a computerized motion capture system and force plates in the floor. Forces between the foot and CDO will be measured using force sensing insoles, and muscle activity data will be collected using surface electromyography. Devices will be mechanically tested, and participant demographic and anthropometric data will be recorded.

ELIGIBILITY:
TIBIAL PILON FRACTURE PARTICIPANTS:

Inclusion Criteria:

* Ages: 18-65
* Sustained unilateral fracture of the tibial pilon within the preceding 5 years
* The fracture has completely healed
* Ability to walk 50 feet without use of an assistive device (cane, crutch, etc.)
* Ability to walk at a slow to moderate pace
* Shoe size between women's 8 and 13.5 or men's 6.5 and 13
* Ability to read and write in English and provide written informed consent
* Individuals with elevated contact stress according to model generated using PedCAT standing CT images (will be answered after completing visit one)

Exclusion Criteria:

* Pain > 6/10 while walking
* Increase in pain during testing of 3/10 or greater
* Neurologic, musculoskeletal (including bilateral fractures) or other condition limiting function of the contralateral extremity
* Medical or psychological condition that would preclude functional testing (ex. moderate or severe brain injury, stroke, heart disease)
* Wounds to the calf that would prevent CDO fitting
* Fractures secondary to neuropathy or severe osteopenia
* Classification as non-ambulatory
* Previous fractures near the tibial pilon on the involved limb
* Surgery on involved limb anticipated in the next 6 months
* Requirement of a knee stabilizing device (i.e. KAFO, KO…) to perform daily activities
* Visual or hearing impairments that limit walking ability or limit the ability to comply with instructions given during testing
* BMI greater than 40
* Pregnancy- Per participant self-report. Due to the expected small number of pregnant individuals and resulting inability to account for its effect on resulting outcomes, participants will be withdrawn from the study.

HEALTHY ABLE-BODIED PARTICIPANTS:

Patient Inclusion Criteria

* Between the ages of 18 and 65
* Shoe size between women's 8 and 13.5 or men's 6.5 and 13
* Healthy individuals without a current complaint of lower extremity pain, spine pain, or medical or neuromusculoskeletal disorders that have limited participation in work or exercise in the last 6 months
* Full active range of motion of the bilateral lower extremities and spine
* Ability to hop without pain
* Ability to perform a full squat without pain
* Ability to read and write in English and provide written informed consent

Patient Exclusion Criteria

* Diagnosed moderate or severe brain injury
* Prior lower extremity injury resulting in surgery or limiting function for greater than 6 weeks
* Diagnosis of a physical or psychological condition that would preclude testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
* Visual or hearing impairment that would interfere with instructions given during testing
* Require an assistive device
* Wounds to the foot or calf that would prevent CDO use
* BMI greater than 40
* Pregnancy - Per participant self-report. Due to the expected small number of pregnant individuals and resulting inability to account for its effect on resulting outcomes, participants will be withdrawn from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: NoCDO, CDOA, CDOB, CDOC: Participants will be evaluated without a CDO, then with CDOA, then with CDOB, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 1: NoCDO, CDOA, CDOC, CDOB: Participants will be evaluated without a CDO, then with CDOA, then with CDOC, then with CDOB.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 1: NoCDO, CDOB, CDOA, CDOC: Participants will be evaluated without a CDO, then with CDOB, then with CDOA, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 1: NoCDO, CDOB, CDOC, CDOA: Participants will be evaluated without a CDO, then with CDOB, then with CDOC, then with CDOA.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 1: NoCDO, CDOC, CDOA, CDOB: Participants will be evaluated without a CDO, then with CDOC, then with CDOA, then with CDOB.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 1: NoCDO, CDOC, CDOB, CDOA: Participants will be evaluated without a CDO, then with CDOC, then with CDOB, then with CDOA.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 2: NoCDO, CDOA, CDOB, CDOC: Participants will be evaluated without a CDO, then with CDOA, then with CDOB, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 2 the design of the CDO proximal cuff was tested with CDOA using a cuff secured with a Chicago screw and Velcro, CDOB using a cuff secured with a ratcheting system (BOA Dial), and CDOC using a cuff consisting of a posterior and an anterior section secured with Velcro.
- Group 2: NoCDO, CDOA, CDOC, CDOB: Participants will be evaluated without a CDO, then with CDOA, then with CDOC, then with CDOB.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 2 the design of the CDO proximal cuff was tested with CDOA using a cuff secured with a Chicago screw and Velcro, CDOB using a cuff secured with a ratcheting system (BOA Dial), and CDOC using a cuff consisting of a posterior and an anterior section secured with Velcro.
- Group 2: NoCDO, CDOB, CDOA, CDOC: Participants will be evaluated without a CDO, then with CDOB, then with CDOA, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 2 the design of the CDO proximal cuff was tested with CDOA using a cuff secured with a Chicago screw and Velcro, CDOB using a cuff secured with a ratcheting system (BOA Dial), and CDOC using a cuff consisting of a posterior and an anterior section secured with Velcro.
- Group 2: NoCDO, CDOB, CDOC, CDOA: Participants will be evaluated without a CDO, then with CDOB, then with CDOC, then with CDOA.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 2 the design of the CDO proximal cuff was tested with CDOA using a cuff secured with a Chicago screw and Velcro, CDOB using a cuff secured with a ratcheting system (BOA Dial), and CDOC using a cuff consisting of a posterior and an anterior section secured with Velcro.
- Group 2: NoCDO, CDOC, CDOA, CDOB: Participants will be evaluated without a CDO, then with CDOC, then with CDOA, then with CDOB.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 2 the design of the CDO proximal cuff was tested with CDOA using a cuff secured with a Chicago screw and Velcro, CDOB using a cuff secured with a ratcheting system (BOA Dial), and CDOC using a cuff consisting of a posterior and an anterior section secured with Velcro.
- Group 2: NoCDO, CDOC, CDOB, CDOA: Participants will be evaluated without a CDO, then with CDOC, then with CDOB, then with CDOA.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 2 the design of the CDO proximal cuff was tested with CDOA using a cuff secured with a Chicago screw and Velcro, CDOB using a cuff secured with a ratcheting system (BOA Dial), and CDOC using a cuff consisting of a posterior and an anterior section secured with Velcro.
- Group 3: NoCDO, CDOA, CDOB, CDOC: Participants will be evaluated without a CDO, then with CDOA, then with CDOB, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 3 the tightness of the CDO proximal cuff was tested with CDOA testing occurring with the cuff tightened to 30N, CDOB testing occurring with the cuff tightened to 50N, and CDOC testing occurring with the cuff tightened to 70N.
- Group 3: NoCDO, CDOA, CDOC, CDOB: Participants will be evaluated without a CDO, then with CDOA, then with CDOC, then with CDOB.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 3 the tightness of the CDO proximal cuff was tested with CDOA testing occurring with the cuff tightened to 30N, CDOB testing occurring with the cuff tightened to 50N, and CDOC testing occurring with the cuff tightened to 70N.
- Group 3: NoCDO, CDOB, CDOA, CDOC: Participants will be evaluated without a CDO, then with CDOB, then with CDOA, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 3 the tightness of the CDO proximal cuff was tested with CDOA testing occurring with the cuff tightened to 30N, CDOB testing occurring with the cuff tightened to 50N, and CDOC testing occurring with the cuff tightened to 70N.
- Group 3: NoCDO, CDOB, CDOC, CDOA: Participants will be evaluated without a CDO, then with CDOB, then with CDOC, then with CDOA.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 3 the tightness of the CDO proximal cuff was tested with CDOA testing occurring with the cuff tightened to 30N, CDOB testing occurring with the cuff tightened to 50N, and CDOC testing occurring with the cuff tightened to 70N.
- Group 3: NoCDO, CDOC, CDOA, CDOB: Participants will be evaluated without a CDO, then with CDOC, then with CDOA, then with CDOB.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 3 the tightness of the CDO proximal cuff was tested with CDOA testing occurring with the cuff tightened to 30N, CDOB testing occurring with the cuff tightened to 50N, and CDOC testing occurring with the cuff tightened to 70N.
- Group 3: NoCDO, CDOC, CDOB, CDOA: Participants will be evaluated without a CDO, then with CDOC, then with CDOB, then with CDOA.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 3 the tightness of the CDO proximal cuff was tested with CDOA testing occurring with the cuff tightened to 30N, CDOB testing occurring with the cuff tightened to 50N, and CDOC testing occurring with the cuff tightened to 70N.
Period: Overall Study
Arm/Group | Group 1: NoCDO, CDOA, CDOB, CDOC | Group 1: NoCDO, CDOA, CDOC, CDOB | Group 1: NoCDO, CDOB, CDOA, CDOC | Group 1: NoCDO, CDOB, CDOC, CDOA | Group 1: NoCDO, CDOC, CDOA, CDOB | Group 1: NoCDO, CDOC, CDOB, CDOA | Group 2: NoCDO, CDOA, CDOB, CDOC | Group 2: NoCDO, CDOA, CDOC, CDOB | Group 2: NoCDO, CDOB, CDOA, CDOC | Group 2: NoCDO, CDOB, CDOC, CDOA | Group 2: NoCDO, CDOC, CDOA, CDOB | Group 2: NoCDO, CDOC, CDOB, CDOA | Group 3: NoCDO, CDOA, CDOB, CDOC | Group 3: NoCDO, CDOA, CDOC, CDOB | Group 3: NoCDO, CDOB, CDOA, CDOC | Group 3: NoCDO, CDOB, CDOC, CDOA | Group 3: NoCDO, CDOC, CDOA, CDOB | Group 3: NoCDO, CDOC, CDOB, CDOA
Started | 1 | 1 | 3 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 2
Completed | 1 | 1 | 3 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Some randomization options (ex. Group 1: NoCDO, CDOB, CDOC, CDOA) had no participants assigned to them, resulting in an overall number of baseline participants equaling zero.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: NoCDO, CDOA, CDOB, CDOC | Group 1: NoCDO, CDOA, CDOC, CDOB | Group 1: NoCDO, CDOB, CDOA, CDOC | Group 1: NoCDO, CDOB, CDOC, CDOA | Group 1: NoCDO, CDOC, CDOA, CDOB | Group 1: NoCDO, CDOC, CDOB, CDOA | Group 2: NoCDO, CDOA, CDOB, CDOC | Group 2: NoCDO, CDOA, CDOC, CDOB | Group 2: NoCDO, CDOB, CDOA, CDOC | Group 2: NoCDO, CDOB, CDOC, CDOA | Group 2: NoCDO, CDOC, CDOA, CDOB | Group 2: NoCDO, CDOC, CDOB, CDOA | Group 3: NoCDO, CDOA, CDOB, CDOC | Group 3: NoCDO, CDOA, CDOC, CDOB | Group 3: NoCDO, CDOB, CDOA, CDOC | Group 3: NoCDO, CDOB, CDOC, CDOA | Group 3: NoCDO, CDOC, CDOA, CDOB | Group 3: NoCDO, CDOC, CDOB, CDOA | Total
Number analyzed (Participants) | 1 | 1 | 3 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 2 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 3 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 2 | 22
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (0.0) | 40.0 (0.0) | 41.0 (11.3) |  | 27.0 (9.9) |  | 35.0 (21.2) | 59.0 (0.0) | 58.0 (0.0) | 39.0 (0.0) |  |  | 56.0 (0.0) | 23.0 (0.0) | 34.5 (3.5) | 26.0 (9.9) | 29.0 (0.0) | 38.5 (16.3) | 38.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 |  | 1 | 0 | 0 | 1 | 1 | 1 |  |  | 0 | 0 | 1 | 2 | 0 | 2 | 9
  Male | 1 | 1 | 3 |  | 1 |  | 2 | 1 | 0 | 0 |  |  | 1 | 1 | 1 | 0 | 1 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 |  | 1 |  | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 1 | 1 | 3 |  | 1 |  | 2 | 2 | 1 | 1 |  |  | 1 | 1 | 1 | 2 | 1 | 2 | 20
  Unknown or Not Reported | 0 | 0 | 0 |  | 0 |  | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0 |  | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 |  | 0 |  | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0 |  | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 |  | 0 |  | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 3 |  | 2 |  | 1 | 2 | 1 | 1 |  |  | 1 | 1 | 2 | 2 | 1 | 2 | 21
  More than one race | 0 | 0 | 0 |  | 0 |  | 0 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 |  | 0 |  | 1 | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Joint Contact Stress Time Exposure (Model Estimated)
Description: Joint contact stress time exposure (MPA-s/gait cycle) was estimated using a participant specific musculoskeletal model. Peak joint contact stress time exposure (MPA-s/gait cycle) acting on the tibia during the gait cycle were reported. Lower peak contact stress time exposure is considered a better outcome.
Time Frame: Baseline
Population: Peak joint contact stress time exposure was only calculated for participants in group 1.
Measure: Mean (Standard Deviation); unit: MPa-s/gait cycle
Groups:
- Group 1: NoCDO; Group 1: CDOA; Group 1: CDOB; Group 1: CDOC: In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 2: NoCDO; Group 2: CDOA; Group 2: CDOB; Group 2: CDOC: In Group 2 the design of the CDO proximal cuff was tested with CDOA using a cuff secured with a Chicago screw and Velcro, CDOB using a cuff secured with a ratcheting system (BOA Dial), and CDOC using a cuff consisting of a posterior and an anterior section secured with Velcro.
- Group 3: NoCDO; Group 3: CDOA; Group 3: CDOB; Group 3: CDOC: In Group 3 the tightness of the CDO proximal cuff was tested with CDOA testing occurring with the cuff tightened to 30N, CDOB testing occurring with the cuff tightened to 50N, and CDOC testing occurring with the cuff tightened to 70N.
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MPa-s/gait cycle | 4.44 (2.80) | 3.97 (3.33) | 4.08 (2.96) | 4.25 (2.94) |  |  |  |  |  |  |  |

2. Primary Outcome: Peak Plantar Force (Total Foot)
Description: Plantar forces normalized to body weight (N/kg) will be measured across the forefoot (100% of sensor) and normalized to participant body weight as they walk.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
N/kg | 11.3 (1.2) | 10.5 (0.8) | 10.7 (0.7) | 10.4 (0.7) | 11.0 (1.3) | 10.6 (0.8) | 10.2 (0.7) | 10.5 (1.0) | 11.0 (0.9) | 10.3 (0.9) | 10.5 (1.2) | 10.6 (1.0)

3. Primary Outcome: Peak Plantar Force (Hindfoot)
Description: Plantar forces normalized to body weight (N/kg) will be measured across the forefoot (proximal 30% of sensor) as participants walk without a CDO and with each CDO.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 7 | 7 | 7 | 9 | 9 | 9 | 9
N/kg | 8.7 (1.2) | 7.2 (0.9) | 7.7 (0.8) | 7.5 (0.9) | 9.2 (2.0) | 8.2 (1.8) | 7.7 (1.8) | 7.8 (2.1) | 8.9 (1.4) | 7.5 (1.0) | 7.6 (1.5) | 7.8 (1.5)

4. Primary Outcome: Peak Plantar Force (Midfoot)
Description: Plantar forces normalized to body weight (N/kg) will be measured across the forefoot (middle 30% of sensor) as participants walk without a CDO and with each CDO.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 7 | 7 | 7 | 9 | 9 | 9 | 9
N/kg | 3.0 (0.7) | 2.8 (0.9) | 3.1 (1.3) | 2.9 (0.5) | 2.5 (0.9) | 1.6 (0.2) | 1.7 (0.4) | 2.0 (0.7) | 2.1 (0.5) | 2.2 (0.7) | 2.3 (0.6) | 2.3 (0.6)

5. Primary Outcome: Peak Plantar Force (Forefoot)
Description: Plantar forces normalized to body weight (N/kg) will be measured across the forefoot (distal 40% of sensor) as participants walk without a CDO and with each CDO.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
N/kg | 9.7 (1.0) | 7.7 (1.3) | 7.7 (0.9) | 7.7 (0.9) | 9.0 (0.6) | 7.1 (1.9) | 6.4 (2.3) | 6.9 (1.5) | 10.3 (0.9) | 7.8 (1.8) | 8.0 (2.0) | 7.9 (2.0)

6. Primary Outcome: Plantar Force Impulse (Total Foot)
Description: Plantar force impulse normalized to body weight (Ns/kg) across the forefoot (100% of sensor) will be calculated using the integral of the force over the stance phase and normalized to participant body weight as they walk.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Ns/kg
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
Ns/kg | 5.8 (0.5) | 5.7 (0.3) | 6.0 (0.3) | 5.7 (0.3) | 5.4 (0.3) | 5.8 (0.3) | 5.7 (0.4) | 5.9 (0.4) | 5.7 (0.4) | 5.8 (0.6) | 5.9 (0.7) | 5.9 (0.7)

7. Primary Outcome: Plantar Force Impulse (Hindfoot)
Description: Plantar force impulse normalized to body weight (Ns/kg) across the forefoot (proximal 30% of sensor) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Ns/kg
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 7 | 7 | 7 | 9 | 9 | 9 | 9
Ns/kg | 2.0 (0.4) | 2.2 (0.5) | 2.5 (0.5) | 2.2 (0.4) | 2.1 (0.4) | 2.6 (0.8) | 2.7 (0.9) | 2.4 (0.8) | 2.1 (0.5) | 2.5 (0.4) | 2.6 (0.7) | 2.7 (0.6)

8. Primary Outcome: Plantar Force Impulse (Midfoot)
Description: Plantar force impulse normalized to body weight (Ns/kg) across the forefoot (middle 30% of sensor) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Ns/kg
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 7 | 7 | 7 | 9 | 9 | 9 | 9
Ns/kg | 1.1 (0.3) | 1.3 (0.4) | 1.3 (0.5) | 1.2 (0.2) | 0.8 (0.3) | 0.6 (0.1) | 0.6 (0.2) | 0.7 (0.2) | 0.7 (0.2) | 1.0 (0.3) | 1.0 (0.2) | 0.9 (0.2)

9. Primary Outcome: Plantar Force Impulse (Forefoot)
Description: Plantar force impulse normalized to body weight (Ns/kg) across the forefoot (distal 40% of sensor) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Ns/kg
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
Ns/kg | 2.7 (0.3) | 2.3 (0.2) | 2.2 (0.2) | 2.3 (0.1) | 2.5 (0.3) | 2.6 (0.7) | 2.4 (0.8) | 2.5 (0.6) | 2.8 (0.5) | 2.3 (0.5) | 2.3 (0.6) | 2.2 (0.6)

10. Primary Outcome: Numerical Pain Rating Scale (Before Performance Measures - 4SST, 5STS)
Description: Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable. Lower values are better as they indicate less pain.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
score on a scale | 0.6 (1.1) | 0.4 (0.8) | 0.4 (0.8) | 0.6 (1.1) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

11. Primary Outcome: Numerical Pain Rating Scale (After Performance Measures - 4SST, 5STS)
Description: as for outcome 10
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
score on a scale | 0.9 (1.2) | 0.4 (0.8) | 0.6 (1.1) | 0.4 (0.8) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.1 (0.3) | 0.0 (0.0) | 0.1 (0.3) | 0.1 (0.3)

12. Primary Outcome: Participant Device Preference (Rank Order NoCDO, CDOA, CDOB, CDOC)
Description: The participant will rank order their preference for their standard of care device (if applicable), No Device, CDO-A, CDO-B, CDO-C on a questionnaire.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: NoCDO, CDOC, CDOB, CDOA: Participants will be evaluated without a CDO, then with CDOA, then with CDOB, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 1: NoCDO, CDOB, CDOC, CDOA: Participants will be evaluated without a CDO, then with CDOA, then with CDOC, then with CDOB.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 1: CDOC, CDOA, CDOB, NoCDO: Participants will be evaluated without a CDO, then with CDOB, then with CDOA, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 1: NoCDO, CDOC, CDOA, CDOB: Participants will be evaluated without a CDO, then with CDOB, then with CDOC, then with CDOA.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 1: CDOC, NoCDO, CDOB, CDOA: Participants will be evaluated without a CDO, then with CDOC, then with CDOA, then with CDOB.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 1: CDOC, CDOA, NoCDO, CDOB: Participants will be evaluated without a CDO, then with CDOC, then with CDOB, then with CDOA.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 1 CDO stiffness was tested with CDOA being the stiffest (7.0(2.1)Nm/deg, CDOB being the moderate stiffness 5.4(1.4)Nm/deg, and CDOC being the least stiff 3.9(1.2)Nm/deg
- Group 2: CDOA, NoCDO, CDOC, CDOB: Participants will be evaluated without a CDO, then with CDOA, then with CDOB, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 2 the design of the CDO proximal cuff was tested with CDOA using a cuff secured with a Chicago screw and Velcro, CDOB using a cuff secured with a ratcheting system (BOA Dial), and CDOC using a cuff consisting of a posterior and an anterior section secured with Velcro.
- Group 2: NoCDO, CDOB, CDOC, CDOA: Participants will be evaluated without a CDO, then with CDOB, then with CDOA, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 2 the design of the CDO proximal cuff was tested with CDOA using a cuff secured with a Chicago screw and Velcro, CDOB using a cuff secured with a ratcheting system (BOA Dial), and CDOC using a cuff consisting of a posterior and an anterior section secured with Velcro.
- Group 2: NoCDO, CDOC, CDOB, CDOA: Participants will be evaluated without a CDO, then with CDOB, then with CDOC, then with CDOA.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 2 the design of the CDO proximal cuff was tested with CDOA using a cuff secured with a Chicago screw and Velcro, CDOB using a cuff secured with a ratcheting system (BOA Dial), and CDOC using a cuff consisting of a posterior and an anterior section secured with Velcro.
- Group 3: NoCDO, CDOB, CDOA, CDOC: Participants will be evaluated without a CDO, then with CDOA, then with CDOC, then with CDOB.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 3 the tightness of the CDO proximal cuff was tested with CDOA testing occurring with the cuff tightened to 30N, CDOB testing occurring with the cuff tightened to 50N, and CDOC testing occurring with the cuff tightened to 70N.
- Group 3: NoCDO, CDOC, CDOB, CDOA: Participants will be evaluated without a CDO, then with CDOB, then with CDOA, then with CDOC.
  Carbon Fiber Custom Dynamic Orthosis (CDO): The CDO will consist of a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  In Group 3 the tightness of the CDO proximal cuff was tested with CDOA testing occurring with the cuff tightened to 30N, CDOB testing occurring with the cuff tightened to 50N, and CDOC testing occurring with the cuff tightened to 70N.
Arm/Group | Group 1: NoCDO, CDOC, CDOB, CDOA | Group 1: NoCDO, CDOB, CDOC, CDOA | Group 1: CDOC, CDOA, CDOB, NoCDO | Group 1: NoCDO, CDOC, CDOA, CDOB | Group 1: CDOC, NoCDO, CDOB, CDOA | Group 1: CDOC, CDOA, NoCDO, CDOB | Group 2: CDOA, NoCDO, CDOC, CDOB | Group 2: NoCDO, CDOA, CDOC, CDOB | Group 2: NoCDO, CDOB, CDOC, CDOA | Group 2: NoCDO, CDOC, CDOB, CDOA | Group 3: NoCDO, CDOA, CDOB, CDOC | Group 3: NoCDO, CDOB, CDOA, CDOC | Group 3: NoCDO, CDOC, CDOB, CDOA | Group 3: NoCDO, CDOB, CDOC, CDOA
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
Participants | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 2 | 2 | 2

13. Primary Outcome: Participant Device Preference (First Preferred Condition)
Description: Participants were asked to rank order their preference for NoCDO, CDO-A, CDO-B, CDO-C on a questionnaire.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
Participants | 4 | 0 | 0 | 3 | 5 | 1 | 0 | 0 | 9 | 0 | 0 | 0

14. Primary Outcome: Participant Device Preference (Second Preferred Condition)
Description: Participants were asked to rank order the testing conditions from the condition they would most prefer to walk in everyday (first preferred) to the condition they would least prefer to walk in everyday (fourth preferred).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
Participants | 1 | 2 | 1 | 3 | 1 | 1 | 1 | 3 | 0 | 3 | 4 | 2

15. Primary Outcome: Participant Device Preference (Third Preferred Condition)
Description: as for outcome 14
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
Participants | 1 | 2 | 3 | 1 | 0 | 0 | 3 | 3 | 0 | 2 | 5 | 2

16. Primary Outcome: Participant Device Preference (Fourth Preferred Condition)
Description: as for outcome 14
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
Participants | 1 | 3 | 3 | 0 | 0 | 4 | 2 | 0 | 0 | 4 | 0 | 5

17. Secondary Outcome: Peak Soleus Muscle Force (Model Estimated)
Description: Peak soleus muscle force (N) during gait was estimated using a participant specific musculoskeletal model.
Time Frame: Baseline
Population: Peak soleus muscle force was only calculate for participants in group 1.
Measure: Mean (Standard Deviation); unit: N
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
N | 2014.4 (408.2) | 1344.8 (754.0) | 1529.6 (479.3) | 1534.5 (487.5) |  |  |  |  |  |  |  |

18. Secondary Outcome: Peak Gastrocnemius Muscle Force (Model Estimated)
Description: Peak gastrocnemius muscle force (N) during gait was estimated using a participant specific musculoskeletal model.
Time Frame: Baseline
Population: Peak gastrocnemius muscle force was only calculated for participants in group 1.
Measure: Mean (Standard Deviation); unit: N
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
N | 1670.3 (328.6) | 1425.4 (559.1) | 1568.0 (464.3) | 1593.4 (426.9) |  |  |  |  |  |  |  |

19. Secondary Outcome: Ankle Range of Motion
Description: Peak ankle dorsiflexion (degrees) during gait.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 7 | 7 | 7 | 9 | 9 | 9 | 9
degree | 17.0 (2.5) | 13.3 (1.9) | 12.9 (1.6) | 13.6 (1.8) | 16.3 (2.5) | 12.3 (1.4) | 12.4 (1.3) | 12.3 (1.4) | 17.1 (3.2) | 13.4 (2.5) | 12.8 (2.6) | 12.6 (2.4)

20. Secondary Outcome: Peak Ankle Moment
Description: Peak ankle plantarflexion moment (Nm/kg) during gait.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 7 | 7 | 7 | 9 | 9 | 9 | 9
Nm/kg | 1.5 (0.1) | 1.5 (0.1) | 1.5 (0.1) | 1.5 (0.2) | 1.4 (0.1) | 1.5 (0.1) | 1.5 (0.1) | 1.5 (0.1) | 1.4 (0.2) | 1.4 (0.2) | 1.4 (0.2) | 1.4 (0.2)

21. Secondary Outcome: Peak Ankle Power
Description: Peak ankle push-off power (W/kg) during gait.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 7 | 7 | 7 | 9 | 9 | 9 | 9
W/kg | 3.0 (0.8) | 1.2 (0.4) | 1.4 (0.5) | 1.6 (0.6) | 2.6 (0.7) | 1.4 (0.2) | 1.2 (0.2) | 1.4 (0.1) | 3.5 (0.6) | 1.5 (0.4) | 1.5 (0.4) | 1.5 (0.4)

22. Secondary Outcome: Four Square Step Test (4SST)
Description: The 4SST (s) is a standardized timed test of balance and agility. One inch pipe is placed on the floor in the shape of a Maltese cross and participants are instructed to begin in the back left quadrant then to move 1) forward, 2) sideways right, 3) backward, then 4) sideways left, then to move in the reverse direction back to the original square.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
seconds | 6.6 (1.7) | 6.6 (1.5) | 6.5 (1.5) | 6.3 (1.4) | 7.1 (2.9) | 7.2 (2.4) | 7.0 (2.2) | 6.7 (2.0) | 6.1 (0.9) | 6.3 (1.1) | 6.4 (1.0) | 6.5 (1.1)

23. Secondary Outcome: Sit to Stand 5 Times (STS5)
Description: STS5 (s) is a well-established timed measure of lower limb muscle strength and power. Participants are instructed to start the test sitting with their arms folded across their chest and with their back against a standard chair. Patients are then instructed to stand up and sit down 5 times as fast as possible, avoiding touching their back to the chair during each repetition. The time to complete all five continuous repetitions is reported.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 9
seconds | 7.9 (2.3) | 8.8 (2.7) | 8.6 (2.5) | 8.4 (2.4) | 7.3 (1.5) | 9.7 (2.4) | 8.8 (1.5) | 8.9 (1.7) | 7.0 (1.3) | 7.5 (1.5) | 7.7 (1.8) | 7.8 (1.6)

24. Secondary Outcome: The Orthotics Prosthetics Users' Survey (OPUS)
Description: Satisfaction with device will be assessed using the Orthotics Prosthetics Users' Survey Satisfaction With Device Score (11-55). Lower scores indicate a better outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 6 | 6 | 9 | 9 | 9
score on a scale | 29.0 (10.9) | 30.3 (8.1) | 31.7 (9.7) | 23.3 (12.6) | 23.8 (13.4) | 26.0 (14.7) | 37.8 (4.0) | 36.3 (3.4) | 36.6 (4.0)

25. Secondary Outcome: Modified Socket Comfort Score (Comfort)
Description: Comfort scores range from 0 = most uncomfortable to 10 = most comfortable. Higher scores are better as they indicate a more comfortable device.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 6 | 6 | 9 | 9 | 9
score on a scale | 6.3 (1.8) | 6.4 (2.0) | 7.6 (1.3) | 7.0 (1.3) | 7.0 (1.4) | 7.7 (0.8) | 7.1 (2.6) | 7.4 (2.2) | 6.7 (2.2)

26. Secondary Outcome: Modified Socket Comfort Score (Smoothness)
Description: Comfort scores range from 0 = least smooth to 10 = most smooth. Higher scores are better as they indicate a smoother rollover with the device.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 6 | 6 | 9 | 9 | 9
score on a scale | 6.1 (1.6) | 5.7 (2.1) | 7.7 (2.0) | 6.5 (2.1) | 6.8 (0.8) | 7.7 (1.4) | 7.7 (1.9) | 7.6 (1.8) | 7.1 (1.9)

27. Other Pre Specified Outcome: Semi-Structured Interview
Description: Semi-structured interviews will also be used to fully capture the patients' perspectives, experience, and opinions associated with the device options they experienced as part of the study.
Time Frame: Baseline
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Center of Pressure Velocity Timing
Description: Timing of peak center of pressure velocity (percent stance) during gait.
Time Frame: Baseline
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Center of Pressure Velocity Magnitude
Description: Magnitude of peak center of pressure velocity (m/s) during gait.
Time Frame: Baseline
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Soleus Muscle Activity (Electromyography)
Description: Electromyography (EMG, % Maximum) of the soleus during gait.
Time Frame: Baseline
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Tibialis Anterior Muscle Activity (Electromyography)
Description: Electromyography (EMG, % Maximum) of theTibialis Anterior during gait.
Time Frame: Baseline
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Medial Gastrocnemius Muscle Activity (Electromyography)
Description: Electromyography (EMG, % Maximum) of the Medial Gastrocnemius during gait.
Time Frame: Baseline
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Rectus Femoris Muscle Activity (Electromyography)
Description: Electromyography (EMG, % Maximum) of the Rectus Femoris during gait.
Time Frame: Baseline
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Vastus Medialis Muscle Activity (Electromyography)
Description: Electromyography (EMG, % Maximum) of the Vastus Medialis during gait.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study participants were asked to indicate any adverse events throughout the duration of each study visit. After completion of the study participants were also asked to call or email the research team if any adverse events related to the study occurred after the study visit (up to ~12 months after the visit).
Arm/Group | Group 1: NoCDO | Group 1: CDOA | Group 1: CDOB | Group 1: CDOC | Group 2: NoCDO | Group 2: CDOA | Group 2: CDOB | Group 2: CDOC | Group 3: NoCDO | Group 3: CDOA | Group 3: CDOB | Group 3: CDOC
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT04562896/Prot_SAP_000.pdf